CLINICAL TRIAL: NCT06528496
Title: N10: Reduced Therapy for High-Risk Neuroblastoma
Brief Title: N10: A Study of Reduced Chemotherapy and Monoclonal Antibody (mAb)-Based Therapy in Children With Neuroblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-144
Record Dates: First submitted 2024-07-22; First posted 2024-07-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: High-risk Neuroblastoma; Neuroblastoma; Childhood Neuroblastoma
Keywords: High-risk neuroblastoma; neuroblastoma; childhood neuroblastoma; N10; Memorial Sloan Kettering Cancer Center; 24-144
MeSH Terms: conditions — Neuroblastoma | interventions — naxitamab; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Cyclophosphamide; Topotecan; Vincristine; Doxorubicin; Ifosfamide; Etoposide; etoposide phosphate; Carboplatin; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Participants with Neuroblastoma (Experimental): Participants will receive 4 cycles of induction chemotherapy followed by a response-based intervention.
  Interventions: Biological: DANYELZA; Biological: Sargramostim; Drug: Cytoxan; Drug: Topotecan; Drug: Vincristine; Drug: Doxorubicin; Drug: Ifosfamide; Drug: Etoposide; Drug: Carboplatin; Drug: Irinotecan; Drug: Temozolomide

INTERVENTIONS:
Biological: DANYELZA — DANYELZA is a humanized monoclonal antibody of the IgG1 subclass
  Other Names: Naxitamab
Biological: Sargramostim — Yeast derived recombinant human Sargramostim (GM-CSF)
  Other Names: granulocyte-macrophage colony-stimulating factor; GM-CSF
Drug: Cytoxan — Cyclophosphamide is an alkylating agent related to nitrogen mustard
  Other Names: Cyclophosphamide
Drug: Topotecan — Topotecan is a topoisomerase I-inhibitor that is a semisynthetic derivative of camptothecin.
Drug: Vincristine — Vincristine is an alkaloid isolated from Vinca rosea Linn (periwinkle).
  Other Names: Oncovin
Drug: Doxorubicin — Doxorubicin is an anthracycline antibiotic
  Other Names: Adriamycin
Drug: Ifosfamide — Ifosfamide is a structural analogue of cyclophosphamide
  Other Names: Isophosphamide
Drug: Etoposide — Etoposide for Injection is available as a 20 mg/mL solution in sterile multiple dose vials (5 mL, 25 mL, or 50 mL each).
  Other Names: VePesid; Etopophos; VP-16
Drug: Carboplatin — Carboplatin is available in 50 mg, 150 mg, 450 mg, and 600 mg vials.
  Other Names: Paraplatin
Drug: Irinotecan — Irinotecan hydrochloride trihydrate (CPT-11) is a topoisomerase I inhibitor
  Other Names: Camptosar
Drug: Temozolomide — Temozolomide is administered intravenously
  Other Names: Temodar

SUMMARY:
The purpose of this study is to find out whether N10 chemotherapy is a safe and effective treatment for children with high-risk neuroblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by histopathology, BM metastases plus high urine catecholamine levels, or positivity in MIBG scan.
* HR-NB, defined as MYCN-amplified stage L2/M/MS at any age and stage M in patients >18 months old.
* No more than one prior cycle of HR-NB chemotherapy
* Age <19 years.
* Signed informed consent indicating awareness of the investigational nature of this treatment.

Exclusion Criteria:

* Severe dysfunction of major organs, i.e., renal, cardiac, hepatic, neurologic, pulmonary, hematologic, or gastrointestinal toxicity >/= to grade 3

  °Organ dysfunction due to direct effects of primary tumor or metastatic disease, or due to paraneoplastic syndromes associated with neuroblastoma, will not be considered in exclusion criteria. Similarly, complications of interventions to control above direct effects (e.g., steroid- induced hyperglycemia or hypertension) will also not be considered in exclusion criteria
* Inability to comply with protocol requirements
* Pregnancy

Ages: 18 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2029-07-22 (Estimated); Study Completion 2029-07-22 (Estimated)

PRIMARY OUTCOMES:
Evaluate participant response | After 2 cycles of mAb-based therapy (each cycle is 21 days)
  To assess the early Complete Response/CR rate in newly-diagnosed HR-NB patients.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org